CLINICAL TRIAL: NCT04813042
Title: The Working Out Dads (WOD) Trial: Comparing the Effectiveness of a Group Peer-Support Intervention (WOD) With Usual Care in Reducing the Mental Health Difficulties of Fathers of Young Children
Brief Title: Determining the Effectiveness of Working Out Dads to Reduce Mental Health Difficulties in Fathers of Young Children
Acronym: WOD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: University of Melbourne (Other); Tweddle Child and Family Health Service (Unknown); Australian National University (Other); La Trobe University (Other); Swinburne University of Technology (Other); Deakin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69411
Record Dates: First submitted 2021-03-10; First posted 2021-03-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-07

CONDITIONS: Mental Health Issue
Keywords: mental health; fathers; men; early fatherhood; peer group intervention
MeSH Terms: conditions — Psychological Well-Being; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: This is a parallel group randomised controlled trial. The treatment (Working Out Dads 6-week group intervention) will be compared to usual care (brief consultation + resources + referral). Randomisation and analyses will be at the level of the individual participant and adjusted for clustering at the level of the WOD group and Local Government Area (LGA) as a stratification variable. For the primary analysis, the model based mean K10 score in each trial arm will be compared at post-intervention and at the 6-month follow-up (primary outcome).
Masking Description: Treatment allocation will be concealed prior to randomisation by the use of a web-based randomisation system. A statistician not directly involved in the analysis of the trial results will prepare the randomisation schedule using permuted block randomisation, stratified by LGA, using a random number generator on a computer. The schedule will be held by the independent statistician and embedded within the web-based data management system.
  Treatment allocation will only be revealed after it has been confirmed that the participant is eligible and enrolled and has completed the baseline questionnaire. REDCap will display the father's assignment for the Project Coordinator, who will notify the father of his treatment assignment and intervention/usual care information by telephone. The treatment allocation in the database will only be visible to the Project Coordinator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Working Out Dads (Experimental): Fathers allocated to the Working Out Dads (WOD) arm will receive the intervention program. WOD is a 6-week manualised program. The weekly 90 minute sessions combine a one hour facilitated discussion by a male facilitator trained in delivery of WOD and a 30-minute gym workout provided by a personal trainer. The group size ranges from 6-10 fathers, with 14 groups running over the study period. The weekly sessions are provided in the evenings, in local gyms or a community setting (e.g., maternal child health centre, local council rooms, local hall, local park, Tweddle Child & Family Health Service).
  Interventions: Behavioral: Working Out Dads
- Usual Care (Active Comparator): Fathers allocated to the Usual Care arm will receive the clinical care typically provided to parents experiencing mental health difficulties by an Early Parenting Centre or community health service. Within 2 weeks of baseline assessment, Usual Care participants will receive a brief psychological consultation from Tweddle's Clinical Manager.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Working Out Dads — The WOD is a manualised group intervention underpinned by solution-focused therapy and social cognitive theories. Psychoeducation about the transition to fatherhood and its potential impacts on wellbeing and family relationships is provided. Fathers are encouraged to share practical ideas for managing stress, revisit previous strategies, validate what they are doing well, and explore solutions.
  The group discussion is followed by a structured group fitness session provided by a personal trainer. This session focuses on body weight exercises, cardio-based activities, stretching, mobility and incidental activity.
  Fathers in the WOD study arm receive 10 weeks of encouraging text messages - one each week during the intervention, and four in the weeks after. These will be sent via the WhatsApp group created for each WOD group. These text messages and the WhatsApp group are designed to facilitate fathers' active engagement with the intervention, and to maintain contact with each other.
  Arms: Working Out Dads
Behavioral: Usual care — The Usual Care arm, also known as 'Talking about being dad' comprises a telephone consultation with a qualified mental health professional. Topics including in this consultation include: (a) discuss family and fathering; (b) health and wellbeing; (c) mental health symptoms and conduct a risk assessment for suicidal ideation; (d) current supports and support needs; (e) provide referral options to telephone support services (PANDA; MensLine); and (f) encourage a general practitioner visit to discuss a mental health care plan.
  Other Names: Talking about being a Dad
  Arms: Usual Care

SUMMARY:
This is an individually randomised trial, where Working Out Dads (WOD) will be delivered as a group intervention. Participants will be randomised to one of two groups: either WOD or usual care.The trial aims to test the effectiveness and cost-effectiveness of WOD, a 6-week week group-based peer support intervention, in reducing fathers' mental health difficulties in early parenthood.

DETAILED DESCRIPTION:
This is an individually randomised trial, where Working Out Dads (WOD) will be delivered as a group intervention.

The primary aim of this study is to test the effectiveness and cost-effectiveness of WOD in reducing fathers' mental health difficulties in early parenthood. A second aim is to identify barriers and facilitators for sustained use and scalability of the WOD program and its adaptation across Victoria and Australia in the future.

Participants will be 280 fathers of young children (0-4 years) who are experiencing mental health difficulties or at risk of poor mental health and suicide. Approximately 140 fathers will be randomised to WOD, and 140 fathers randomised to usual care.

Fathers will be recruited from four Victorian Local Government Areas (LGAs): Wyndham, Whittlesea, Geelong, and Ballarat. Within these sites, fathers will be recruited through maternal and child health, medical and family support services.

Data will be collected via self-report surveys at baseline, 10 weeks, 24 weeks, 18 months, and 3 years. The assessment at 24 weeks will also include a telephone interview with a researcher (blinded) to assess mental health. In August 2022, an optional 72-week follow-up was added to the study design.

Participants will be randomised in a 1:1 ratio to the two treatment arms. A statistician not directly involved in the analysis of the trial results will prepare the randomisation schedule using permuted block randomisation, stratified by LGA, using a random number generator on a computer. The schedule will be held by the independent statistician and embedded within the web-based data management system.

Treatment arms:

Intervention condition - WOD: Fathers will attend a WOD group within approximately two weeks of randomisation and within four weeks of baseline assessment. WOD is a 6-week group-based peer support intervention. WOD's weekly sessions consists of 1-hour group discussion focused on common challenges and risk factors for poor mental health in early fatherhood, followed by a 30-minute group exercise session. Fathers in the WOD intervention condition will also have access to online resources and a father-managed WhatsApp group.

Usual care condition: Fathers will receive the clinical care typically provided by an early parenting or community health service to parents experiencing mental health difficulties. Within two weeks of baseline assessment, Tweddle's Clinical Manager will conduct a brief telephone consultation to: (a) enquire about mental health symptoms and conduct a risk assessment for suicidal ideation; (b) provide referral options to telephone support services (e.g., PANDA, MensLine); and (c) encourage visiting a general practitioner to discuss accessing a mental health care plan.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18 years or older
* Be biological or step-father, or male caregiver of a child aged 0-4 years
* Be in regular weekly contact with the child, even if non-resident parent
* Be sufficiently fluent in English to complete surveys and participate in the intervention
* Have mental health difficulties above the symptomatic cut-point (score of 20+) on the K10.

AND/OR

• Have at least two risk factors for poor mental health/suicide including: (a) history of mental health difficulties; (b) relationship difficulties; (c) high work-related stress; (d) unemployment; or (e) have a child with sleep difficulties, a disability, chronic illness or other special health care need.

Exclusion Criteria:

* Has a severe mental health disorder - self reported psychosis, substance use dependency, prescribed anti-psychotic medication that may require more intensive mental health interventions and treatment
* Has an overt indicator of family violence - self-reported intervention order or court case for family violence
* Has child protection service involvement

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 293 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Kessler Psychological Distress Scale, mean difference in total scale scores between the Working Out Dads and Usual Care arms | post intervention at week 24
  The 10-item Kessler Psychological Distress Scale (K10) assesses depressive and anxiety symptoms in the last 4 weeks. Scores range from 10-50 with higher scores indicating greater levels of psychological distress. Rationale: The K10 is widely used in clinical trials for common mental health disorders, and is consistent with a transdiagnostic approach proposing a common set of psychological distress symptoms underlie mood and anxiety disorders.

SECONDARY OUTCOMES:
The Mini International Neuropsychiatric Interview mean difference in proportion of depressive, suicidal, and anxiety mental health disorders between Working Out Dads and Usual Care arms | post intervention at week 24
  The Mini International Neuropsychiatric Interview (MINI) will be used to determine clinically significant depressive, suicidal or anxiety mental health disorders. Administered via telephone by trained staff, this 15-minute structured diagnostic interview assesses 17 common DSM-5 and ICD-10 psychiatric disorders. It is well validated for use in clinical trials and epidemiological studies. In this prevention trial, we predict a higher proportion of fathers in the usual care arm (vs. the intervention arm) will have ongoing or emerging clinically significant depressive, suicidal or anxiety mental health disorders by 6 months
The Depression Anxiety Stress Scale-21mean difference scale scores between Working Out Dads and Usual Care arms | post intervention at week 10
  The Depression Anxiety Stress Scale-21 (DASS-21) assesses symptoms of depression, anxiety, and stress in the past week (21 items). Scores on each scale range from 0-42 with higher scores indicating a greater severity of symptoms.Clinical ranges are available. Excellent reliability and validity has been demonstrated in Australian population-based samples. The DASS-21 is routinely used by early parenting services.
The Depression Anxiety Stress Scale-21 mean difference scale scores between the Working Out Dads and Usual Care arms | post intervention at week 24
  The Depression Anxiety Stress Scale-21 (DASS-21) assesses symptoms of depression, anxiety, and stress in the past week (21 items). Scores on each scale range from 0-42 with higher scores indicating a greater severity of symptoms. Clinical ranges are available. Excellent reliability and validity has been demonstrated in Australian population-based samples. The DASS-21 is routinely used by early parenting services.
The Depression Anxiety Stress Scale-21 mean difference scale scores between the Working Out Dads and Usual Care arms | post intervention at week 72
  The Depression Anxiety Stress Scale-21 (DASS-21) assesses symptoms of depression, anxiety, and stress in the past week (21 items). Scores on each scale range from 0-42 with higher scores indicating a greater severity of symptoms. Clinical ranges are available. Excellent reliability and validity has been demonstrated in Australian population-based samples. The DASS-21 is routinely used by early parenting services.
The Suicidal Ideation Attributes Scale mean difference in total scale scores between the Working Out Dads and Usual Care arms | post intervention at week 10
  The Suicidal Ideation Attributes Scale is a 5-item screener for the presence and severity of suicidal thoughts in the last month based on frequency, controllability, closeness to attempt, level of distress, and impact on daily functioning. Scores range from 0-50 with higher scores indicating a greater severity of suicidal ideation. Any ideation is indicative of risk for suicidal behaviour; scores >21 indicate high risk. Online administration has been validated (N=1352 Australian adults), and it has excellent reliability (Cronbach α=0.91) and validity.
The Suicidal Ideation Attributes Scale mean difference in total scale scores between the Working Out Dads and Usual Care arms | post intervention at week 24
  The Suicidal Ideation Attributes Scale is a 5-item screener for the presence and severity of suicidal thoughts in the last month based on frequency, controllability, closeness to attempt, level of distress, and impact on daily functioning. Scores range from 0-50 with higher scores indicating a greater severity of suicidal ideation. Any ideation is indicative of risk for suicidal behaviour; scores >21 indicate high risk. Online administration has been validated (N=1352 Australian adults), and it has excellent reliability (Cronbach α=0.91) and validity.
The Suicidal Ideation Attributes Scale mean difference in total scale scores between the Working Out Dads and Usual Care arms | post intervention at week 72
  The Suicidal Ideation Attributes Scale is a 5-item screener for the presence and severity of suicidal thoughts in the last month based on frequency, controllability, closeness to attempt, level of distress, and impact on daily functioning. Scores range from 0-50 with higher scores indicating a greater severity of suicidal ideation. Any ideation is indicative of risk for suicidal behaviour; scores >21 indicate high risk. Online administration has been validated (N=1352 Australian adults), and it has excellent reliability (Cronbach α=0.91) and validity.
The Medical Outcomes Study-Social Support Survey mean difference in total scale scores between the Working Out Dads and Usual Care arms | post intervention at week 24
  The Medical Outcomes Study-Social Support Survey (MSSS). The 14 items assess tangible, emotional, affective and positive support. Scores range from 14-70 with higher scores indicating greater levels of perceived social support. Excellent reliability (Cronbach's α=0.88) and validity have been established.
The Medical Outcomes Study-Social Support Survey mean difference in total scale scores between the Working Out Dads and Usual Care arms | post intervention at week 10
  The Medical Outcomes Study-Social Support Survey (MSSS). The 14 items assess tangible, emotional, affective and positive support. Scores range from 14-70 with higher scores indicating greater levels of perceived social support. Excellent reliability (Cronbach's α=0.88) and validity have been established.
The Medical Outcomes Study-Social Support Survey mean difference in total scale scores between the Working Out Dads and Usual Care arms | post intervention at week 72
  The Medical Outcomes Study-Social Support Survey (MSSS). The 14 items assess tangible, emotional, affective and positive support. Scores range from 14-70 with higher scores indicating greater levels of perceived social support. Excellent reliability (Cronbach's α=0.88) and validity have been established.
Perceived Need for Care Questionnaire (modified version), mean difference in proportion with unmet need between the Working Out Dads and Usual Care arms | post intervention at week 24
  A modified version of the Perceived Need for Care Questionnaire will be used to ask fathers if they needed mental health care but could not access (same time period). Fathers will be as either as either 0= having no unmet need, or 1= having unmet needs.
Perceived Need for Care Questionnaire (modified version), mean difference in proportion with unmet need between the Working Out Dads and Usual Care arms | post intervention at week 72
  A modified version of the Perceived Need for Care Questionnaire will be used to ask fathers if they needed mental health care but could not access (same time period). Fathers will be as either as either 0= having no unmet need, or 1= having unmet needs.
The Revised Attitudes Towards Seeking Professional Psychological Help Scale mean difference in total scale scores between the Working Out Dads and Usual Care arms | post intervention at week 24
  The 10-item Revised Attitudes Towards Seeking Professional Psychological Help Scale.Scores range from 0-30 with higher scores indicating a more positive attitude towards help-seeking. Excellent reliability has been established in Australian samples (Cronbach's α=0.77).
The Karitane Parenting Confidence Scale mean difference in total scale scores between the Working Out Dads and Usual Care arms | post intervention at week 24
  The Karitane Parenting Confidence Scale (KPCS) is a 15-item measure that assesses parents' perceived parenting self-efficacy or sense of competence in their parenting abilities. Scores range from 0-45 with higher scores indicating a greater level of parenting self-efficacy. The scale has documented excellent internal consistency, test-retest reliability, convergent and discriminant validity with mothers of young children.
The Child-Parent Relationship Scale- short form mean difference in total scale scores between the Working Out Dads and Usual Care arms | post intervention at week 24
  The Child-Parent Relationship Scale- short form (CPRS) is a 15-item measure which assess parents' perceptions of their relationship with their child. The measure is comprised of two subscales: closeness and conflict. Scores on the Conflict subscale range between 8-40 with higher scores indicating greater levels of perceived parent-child conflict. Scores on the closeness subscale range between 7-35 with higher scores indicating greater parent-child closeness.
Health Service Use cost, mean difference in cost of healthcare use between the Working Out Dads and Usual Care arms | post intervention at week 24
  Service use will be assessed by self-reported cost of healthcare services accessed (prior to baseline and during the study period) and by examination of Medicare data. Higher cost will indicate a greater expense of health care use.
Health Service Use, mean difference in number of healthcare use between the Working Out Dads and Usual Care arms | post intervention at week 24
  Service use will be assessed by self-reported number of healthcare services accessed (prior to baseline and during the study period) and by examination of Medicare data. Higher numbers will indicate a higher frequency of health care use.
Health Service Use, mean difference in number of healthcare use between the Working Out Dads and Usual Care arms | post intervention at week 72
  Service use will be assessed by self-reported number of healthcare services accessed (prior to baseline and during the study period) and by examination of Medicare data. Higher numbers will indicate a higher frequency of health care use.
The Assessment of Quality of Life 8 dimension, mean difference in preference weighted health related quality of life utility scores between the Working Out Dads and Usual Care arms | post intervention at week 24
  The Assessment of Quality of Life 8 dimension (AQoL-8D), is a validated tool assessing quality of life impacts in the economic evaluation. Australian population normative data are available and will be used to determine preference weighted health related quality of life utility scores ranging from 0-1 with higher scores indicating higher quality of life. The AQoL-8D is particularly suited to measuring mental health aspects of quality of life.
The Assessment of Quality of Life 8 dimension, mean difference in preference weighted health related quality of life utility scores between the Working Out Dads and Usual Care arms | post intervention at week 72
  The Assessment of Quality of Life 8 dimension (AQoL-8D), is a validated tool assessing quality of life impacts in the economic evaluation. Australian population normative data are available and will be used to determine preference weighted health related quality of life utility scores ranging from 0-1 with higher scores indicating higher quality of life. The AQoL-8D is particularly suited to measuring mental health aspects of quality of life.
The Kessler Psychological Distress Scale mean difference in total scale scores between the Working Out Dads and Usual Care arms | post intervention at week 10
  The 10-item Kessler Psychological Distress Scale (K10). assesses depressive and anxiety symptoms in the last 4 weeks. Scores range from 10-50 with higher scores indicating greater levels of psychological distress. Rationale: The K10 is widely used in clinical trials for common mental health disorders, and is consistent with a transdiagnostic approach proposing a common set of psychological distress symptoms underlie mood and anxiety disorders.
The Kessler Psychological Distress Scale mean difference in total scale scores between the Working Out Dads and Usual Care arms | post intervention at week 72
  The 10-item Kessler Psychological Distress Scale (K10). assesses depressive and anxiety symptoms in the last 4 weeks. Scores range from 10-50 with higher scores indicating greater levels of psychological distress. Rationale: The K10 is widely used in clinical trials for common mental health disorders, and is consistent with a transdiagnostic approach proposing a common set of psychological distress symptoms underlie mood and anxiety disorders.
Health behaviours mean differences in summed scores between the Working Out Dads and Usual Care arms | post intervention at week 72
  Questions related to alcohol use and physical activity from the AUDIT-C and Active Australia Study, respectively, have been included. Seven study designed items have been developed to ask fathers about the extent to which they are engaging in positive health behaviours (e.g., had enough rest and sleep, exercised regularly, had time to self, spent time with family, friends, and partner).
Me as a Parent Scale mean difference in total scale scores between the Working Out Dads and Usual Care arms. | post intervention at week 72
  The Me as a Parent Scale (MaaPS) is a 16-item scale assessing parent beliefs about self-efficacy, personal agency, self-management and self-sufficiency.
Child-Parent Relationhip Scale mean difference in total scale scores between the Working Out Dads and Usual Care arms. | post intervention at week 72
  The Child-Parent Relationship Scale- short form (CPRS)[39] is a 15-item measure which assess parents' perceptions of their relationship with their child.
Parenting Warmth, hostility and engagement in home learning activities- mean difference in total summed scores between the Working Out Dads and Usual Care arms. | post intervention at week 72
  Parenting hostility will be assessed using four adapted items from the Early Childhood Longitudinal Study of Children. Fathers will rate how often they engage in hostile behaviours during interactions with their child. Parenting warmth will be assessed using a modified six-item subscale from the Child Rearing Questionnaire. Fathers will indicate how often they feel close to and express affection toward their child. Parental Involvement Scale is a five-item scale taken from the Growing Up in Australia: Longitudinal Study of Australian Children assessing the frequency in which parents have done the following activities with their child: read from a book, told a story (not from a book), played with toys/games indoors (e.g., board/card games), involved them in everyday activities at home (e.g., cooking/caring for pets), and played a game outdoors or exercise together (e.g., walking, swimming).
Uptake of father specific supports and/or activities- mean difference in number of activities taken up between the Working Out Dads and Usual Care arms. | post intervention at week 72
  Study specific questions have been developed to ask fathers about what activities (e.g., joined a fathers' group, stayed in contact with other fathers) they have engaged in since participating in WOD or usual care.
The Depression Anxiety Stress Scale-21 mean difference scale scores between the Working Out Dads and Usual Care arms | post intervention at 156 weeks (3 years)
  The Depression Anxiety Stress Scale-21 (DASS-21) assesses symptoms of depression, anxiety, and stress in the past week (21 items). Scores on each scale range from 0-42 with higher scores indicating a greater severity of symptoms. Clinical ranges are available. Excellent reliability and validity has been demonstrated in Australian population-based samples. The DASS-21 is routinely used by early parenting services.
The Suicidal Ideation Attributes Scale mean difference in total scale scores between the Working Out Dads and Usual Care arms | post intervention at week 156 (3 years)
  The Suicidal Ideation Attributes Scale is a 5-item screener for the presence and severity of suicidal thoughts in the last month based on frequency, controllability, closeness to attempt, level of distress, and impact on daily functioning. Scores range from 0-50 with higher scores indicating a greater severity of suicidal ideation. Any ideation is indicative of risk for suicidal behaviour; scores >21 indicate high risk. Online administration has been validated (N=1352 Australian adults), and it has excellent reliability (Cronbach α=0.91) and validity.
The Medical Outcomes Study-Social Support Survey mean difference in total scale scores between the Working Out Dads and Usual Care arms | post intervention at week 156 (3 years)
  The Medical Outcomes Study-Social Support Survey (MSSS). The 14 items assess tangible, emotional, affective and positive support. Scores range from 14-70 with higher scores indicating greater levels of perceived social support. Excellent reliability (Cronbach's α=0.88) and validity have been established.
Perceived Need for Care Questionnaire (modified version), mean difference in proportion with unmet need between the Working Out Dads and Usual Care arms | post intervention at week 156 (3 years)
  A modified version of the Perceived Need for Care Questionnaire will be used to ask fathers if they needed mental health care but could not access (same time period). Fathers will be as either as either 0= having no unmet need, or 1= having unmet needs.
The Child-Parent Relationship Scale- short form mean difference in total scale scores between the Working Out Dads and Usual Care arms | post intervention at week 156 (3 years)
  The Child-Parent Relationship Scale- short form (CPRS) is a 15-item measure which assess parents' perceptions of their relationship with their child. The measure is comprised of two subscales: closeness and conflict. Scores on the Conflict subscale range between 8-40 with higher scores indicating greater levels of perceived parent-child conflict. Scores on the closeness subscale range between 7-35 with higher scores indicating greater parent-child closeness.
Health Service Use, mean difference in number of healthcare use between the Working Out Dads and Usual Care arms | post intervention at week 156 (3 years)
  Service use will be assessed by self-reported number of healthcare services accessed (prior to baseline and during the study period). An adapted reduced number if items will be used for the 3 year follow up. Higher numbers will indicate a higher frequency of health care use.
The Kessler Psychological Distress Scale mean difference in total scale scores between the Working Out Dads and Usual Care arms | post intervention at week 156 (3 years)
  The 10-item Kessler Psychological Distress Scale (K10). assesses depressive and anxiety symptoms in the last 4 weeks. Scores range from 10-50 with higher scores indicating greater levels of psychological distress. Rationale: The K10 is widely used in clinical trials for common mental health disorders, and is consistent with a transdiagnostic approach proposing a common set of psychological distress symptoms underlie mood and anxiety disorders.
Me as a Parent Scale mean difference in total scale scores between the Working Out Dads and Usual Care arms. | post intervention at week 156 (3 years)
  The Me as a Parent Scale (MaaPS) is a 16-item scale assessing parent beliefs about self-efficacy, personal agency, self-management and self-sufficiency.
Parenting Warmth, hostility and engagement in home learning activities- mean difference in total summed scores between the Working Out Dads and Usual Care arms. | post intervention at week 156 (3 years)
  Parenting hostility will be assessed using four adapted items from the Early Childhood Longitudinal Study of Children. Fathers will rate how often they engage in hostile behaviours during interactions with their child. Parenting warmth will be assessed using a modified six-item subscale from the Child Rearing Questionnaire. Fathers will indicate how often they feel close to and express affection toward their child. Parental Involvement Scale is a five-item scale taken from the Growing Up in Australia: Longitudinal Study of Australian Children assessing the frequency in which parents have done the following activities with their child: read from a book, told a story (not from a book), played with toys/games indoors (e.g., board/card games), involved them in everyday activities at home (e.g., cooking/caring for pets), and played a game outdoors or exercise together (e.g., walking, swimming).
Uptake of father specific supports and/or activities- mean difference in number of activities taken up between the Working Out Dads and Usual Care arms. | post intervention at week 156 (3 years)
  Study specific questions have been developed to ask fathers about what activities (e.g., joined a fathers' group, stayed in contact with other fathers) they have engaged in since participating in WOD or usual care.
Perceived burdensomeness and thwarted belongingness difference in mean item response scores between the Working Out Dads and Usual Care arms. | post intervention at week156 (3 years)
  The Interpersonal Needs Questionnaire (INQ) (45) is a 15-item measure that assesses perceived burdensomeness (6 items) and thwarted belongingness (9 items), constructs that are proximal causes of desire for suicide. Participants rate items such as "These days the people in my life would be better off if I were gone" on a seven-point scale ranging from 1 "Not at all true for me", through 4 "Somewhat true for me", to 7 "Very true for me". Items are scored as a mean item response with higher scores indicating higher perceived burdensomeness and thwarted belongingness. This measure has been well validated for use in Western populations and has demonstrated good internal consistency, and construct, factorial, and convergent validity. (45)
professional help-seeking attitudes- mean difference in total scale scores between the Working Out Dads and Usual Care arms | post intervention at week 156 (3 years)
  The Barriers to Help Seeking Scale (BHSS)[33]. The 31-items measure men's perceived barriers to help-seeking for a wellbeing problem. The scale comprises of five subscales: (a) Need for Control and Self-reliance; (b) Minimizing Problems and Resignation; (c) Concrete Barriers and Distrust of Caregivers; (d) Privacy; and (e) Emotional Control. Good construct validity for subscales has been reported along the validity between BHHS and other measures of gender role conflict and attitudes to help-seeking.
professional help-seeking attitudes- mean difference in total scale scores between the Working Out Dads and Usual Care arms | post intervention at week 24 weeks
  The Barriers to Help Seeking Scale (BHSS)[33]. The 31-items measure men's perceived barriers to help-seeking for a wellbeing problem. The scale comprises of five subscales: (a) Need for Control and Self-reliance; (b) Minimizing Problems and Resignation; (c) Concrete Barriers and Distrust of Caregivers; (d) Privacy; and (e) Emotional Control. Good construct validity for subscales has been reported along the validity between BHHS and other measures of gender role conflict and attitudes to help-seeking.
Co-parenting. The Coparenting Relationship Scale, mean difference in subscale scores between WODand the Usual careintervention arms. | 156 - weeks post randomisation - (3 years)
  The Coparenting Relationship Scale consists of 35 items (e.g., my co-parent asks my opinion on issues related to parenting, my co-parent has lots of patience with our child, my relationship with my co-parent is stronger now than before we had a child), comprising seven subscales (Coparenting Agreement, Coparenting Closesness, Exposure to Conflict, Coparenting Support, Coparenting Undermining, Endorse Co-parent Parenting, and Division of Labor). Each item is rated on a 7-point scale, ranging from 0=Not true of us/Never to 6=Very true of us/Often. Particular items are reverse scored, and then summed. The scale is ideal for examining the role of coparenting in diverse family contexts. The subscales have excellent internal reliability with parent populations in the US and Australia.
Interparental conflict. mean difference in total scale scores on the Co-parental Communication Scale between the Working Out Dads and Usual Care arms | post intervention at week 156 (3 years)
  IPC will be assessed using a subscale from the Co-parental Communication Scale used in the Longitudinal Study of Australian Children. This scale consists of five items assessing how often parents engage in verbal conflict (e.g. 'How often do you argue?') and one item assessing how often they engage in physical conflict (e.g. 'How often do you have arguments with your partner that end up with people pushing, hitting, kicking or shoving?'). The items are rated on a 5-point scale from 1 = never to 5 = always. Items scores were summed, with higher scores indicating more frequent IPC. The scale has excellent reliability and validity in Australian father populations .
Work to family conflict mean difference in total scores across 4 adapted items between the Working Out Dads and Usual Care arms | post intervention at week 156 (3 years)
  A 4-item adaptation of the scales authored by Marshall and Barnett will assess employment-related constraints on family life and parenting (e.g., 'Because of my work responsibilities, I have missed out on home or family activities that I would like to take part in) and constraints from family responsibilities that affect employment (e.g. 'Because of my family responsibilities, my work time is less enjoyable and more pressured). The items are rated on a 5 point scale ranging from 1 = strongly disagree to 5 = strongly agree, creating a total scale score with higher scores indicating more work-family conflict. The scale has excellent internal reliability in Australian parent populations.
Total difficulticulties mean difference in total scores between the Working Out Dads and Usual Care arms | post intervention at week 156 (3 years)
  The Strengths and Difficulties Questionnaire Parent version is a widely used tool designed to assess psychological adjustment in children. The measure consists of 25-items divided into five subscales: emotional symptoms, conduct problems, hyperactivity-inattention, peer problems and prosocial behaviour. The first four of these 5-item subscales can be totaled to provide a total difficulties score with higher scores indicating more difficulty. This measure has been extensively validated, including in Australian populations and has demonstrated strong internal reliability across subscales, as well as sound internal and external validity.
positive health behaviours mean difference in total scores between the Working Out Dads and Usual Care arms | post intervention at week 156 (3 years)
  Questions related to alcohol use and physical activity from the AUDIT-C and Active Australia Study, respectively, have been included. Seven study designed items have been developed to ask fathers about the extent to which they are engaging in positive health behaviours (e.g., had enough rest and sleep, exercised regularly, had time to self, spent time with family, friends, and partner). An open-ended question about self-care has also been included.
Difference in occurance of self-harm ideation or behaviour between the Working Out Dads and Usual Care arms | post intervention at week 156 (3 years)
  Two items adapted from LSAC study derived measures will be asked to assess whether participants have either thought about, or intentionally hurt themselves during the past 12 months. Participants respond with either yes or no to both items
Difference in occurance of lietime suicide attempt between the Working Out Dads and Usual Care arms | post intervention at week 156 (3 years)
  Participants will be asked if they have ever made a suicide attempt during their lifetime using a single item from Ten to Men

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Giallo, PhD, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Murdoch Children's Research Institute, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for analysis of the WOD Trial will be available for six months after publication of the primary outcome. The study protocol, data dictionary and analysis plan will also be made available. Medicare and Pharmaseutical Benefits Scheme data will not be available. The de-identified data set will only be made available to researchers from a recognised research institute: (i) who sign a data access agreement accepting MCRI's conditions for access and appropriate acknowledgement, (ii) whose proposed use and analysis plan has been approved by the Sponsor Investigator and the Trial Steering Committee, and (iii) whose proposed use has been reviewed and accepted by the Royal Children's Hospital Human Research Ethics Committee.
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after publication of primary outcome
Access Criteria: (1) Recognised research institute, (2) data access agreement, (3), proposed use approved by Sponsor Investigator and Trial Steering Committee, and (4) proposed use reviewed and accepted by human research ethics committee.

REFERENCES:
- [Derived] Giallo R, Seymour M, Fogarty A, Hosking C, Williams LA, Cooklin A, Grobler A, Ride J, Leach L, Oldenburg B, Wood C, Borschmann R, O'Brien J, Evans K, Treyvaud K, Garfield C, Brown S, Nicholson J. Working out dads (WOD): a study protocol for a randomised controlled trial of a group-based peer support intervention for men experiencing mental health difficulties in early fatherhood. BMC Psychiatry. 2022 Feb 12;22(1):111. doi: 10.1186/s12888-022-03698-5. PMID 35151305